CLINICAL TRIAL: NCT00068783
Title: A Phase II Trial of STI-571/Imatinib (Gleevec®) (NSC-716051) in Neuroendocrine Carcinoma of the Skin (Merkel Cell Carcinoma)
Brief Title: S0331: Imatinib Mesylate in Treating Patients With Metastatic or Unresectable Merkel Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03182; S0331; U10CA032102 (NIH); CDR0000328120 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Neuroendocrine Carcinoma of the Skin; Stage II Neuroendocrine Carcinoma of the Skin; Stage III Neuroendocrine Carcinoma of the Skin
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (Experimental): Patients receive oral imatinib mesylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or symptomatic deterioration.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well imatinib mesylate works in treating patients with metastatic or unresectable Merkel cell cancer. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of a Southwest Oncology Group Phase II trial or oral STI-571/imatinib (Gleevec) administered to patients with metastatic or unresectable Merkel cell carcinoma.

II. To evaluate the objective response probability (confirmed and unconfirmed complete and partial responses) of oral STI-571/imatinib (Gleevec) administered to patients with metastatic or unresectable Merkel cell carcinoma.

III. To assess qualitative and quantitative toxicities of oral STI-581/imatinib (Gleevec) administered to patients with metastatic or unresectable Merkel cell carcinoma.

IV. To analyze tumor samples for activating mutations of STI-571/imatinib-sensitive kinases (KIT, PDGFRA, PDGFRB) by denaturing HPLC and direct DNA sequencing.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or symptomatic deterioration.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a biopsy-proven diagnosis of Merkel Cell Carcinoma (Cutaneous Neuroendocrine Carcinoma) that is distantly metastatic or unresectable

  * Tumors must beet BOTH of the following criteria:

    * The primary must be of skin origin; (patients with unknown primary are not eligible)
    * All patients must have immunohistochemical staining with c-kit (CD117) expression by tumor documented by DAKO, Benchmark, or similar staining kit
* The institution must plan to submit materials for pathology review

  * NOTE: Submission of additional specimens is strongly encouraged
* Patients must have measurable disease; all measurable lesions must be assessed (by physical examination, CT or MRI scan or plain X-ray) within 28 days prior to registration; tests to assess non-measurable disease must be performed within 42 days prior to registration
* Patients with symptomatic, unstable or untreated brain metastases are not eligible; previous treatment must have been completed at least 28 days prior to registration
* Patients must have a Zubrod performance status of 0-2
* Patients must not have received radiotherapy, chemotherapy, biologic therapy or any other investigational drug for any reason within 28 days prior to registration; all toxicities from prior treatment must have been resolved (in the opinion of the treating investigator); patients whose only disease is within a previous radiation therapy port must demonstrate clearly progressive disease prior to registration; patients must have resolution of all toxicities from any prior therapy to =< grade 1 (CTCAE version 3.0); patients must not have had a major surgery (e.g., large chest and abdominal incisions, major soft tissue resections) within 14 days prior to registration
* Serum bilirubin =< 3 x the institutional upper limit of normal (including those with hepatic metastases)
* SGOT or SGPT =< 2.5 x the institutional upper limit of normal (or =< 5 x the institutional upper limit of normal if hepatic metastases is present)
* Serum creatinine =< 1.5 x the institutional upper limit of normal
* ANC >= 1,000/ul
* Platelet count >= 100,000/ul
* Hemoglobin >= 9 gm/dl (this may be achieved by transfusion if needed)
* Patient must not have class 3/4 cardiac problems as defined by the New York Heart Association criteria (e.g., congestive heart failure, myocardial infarction within 2 months of study)
* Patient must not have a sever and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, or active uncontrolled infection, e.g., HIV)
* Patients must not be pregnant or nursing; for women of reproductive potential, a negative serum pregnancy test must be done within 7 days prior to registration; post-menopausal women who have not had their ovaries removed must be amenorrheic for at least 12 months to be considered of non-childbearing potential; patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug

  * NOTE: oral contraceptives may interact with the study drug and should be used with caution
* Patients must not be taking therapeutic doses of Coumadin (warfarin) as anticoagulation at the time of registration; patients requiring therapeutic anticoagulation may use low molecular weight heparin (e.g., Lovenox) or other agents, and mini-dose Coumadin (1 mg po QD) as prophylaxis is allowed
* If day 7, 14, or 42 falls on a weekend or holiday, the limit may be extended to the next working day

  * In calculating days of tests and measurements, the day a test or measurement is dose is considered day 0; therefore, if a test is done on a Monday, the Monday two weeks later would be considered day 14; this allows for efficient patient scheduling without exceeding the guidelines
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-10; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response probability | Up to 4 years

SECONDARY OUTCOMES:
Toxicity rates | Up to 4 years
  Estimated with 95% confidence interval.
Mutation rate for KIT | Baseline
  Estimated with 95% confidence interval.
Mutation rate for PDGFRA | Baseline
  Estimated with 95% confidence interval.
Mutation rate for PDGFRB | Baseline
  Estimated with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Samlowski, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States